CLINICAL TRIAL: NCT06519591
Title: Systemic Application of Cadonilimab, LM-302, and S-1 Combined With Intraperitoneal Infusion of Paclitaxel for the Treatment of Claudin 18.2-positive Gastric Cancer With Peritoneal Metastasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, YANGZHONGYIN, Doctor, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRAGON-12
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer Stage IV; Peritoneal Metastases
Keywords: Gastric cancer; Peritoneal metastasis; Cadonilimab; Claudin 18.2; Paclitaxel
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Cadonilimab 10mg/kg, LM-302 2.0mg/kg intravenous (IV) infusion on day 1, paclitaxel 20 mg/m2 intraperitoneal infusion on Days 1 and 8 plus oral S-1 80 mg/m2 for 14 consecutive days every 3 weeks.
  Interventions: Drug: Cadonilimab, LM-302, S-1, paclitaxel

INTERVENTIONS:
Drug: Cadonilimab, LM-302, S-1, paclitaxel — Cadonilimab 10mg/kg, LM-302 2.0mg/kg intravenous (IV) infusion on day 1, paclitaxel 20 mg/m2 intraperitoneal infusion on Days 1 and 8 plus oral S-1 80 mg/m2 for 14 consecutive days every 3 weeks.

SUMMARY:
In this phase 2 study, we combined Cadonilimab, LM-302, and S-1 combined with intraperitoneal infusion of paclitaxel as regimen to treat gastric cancer patients with peritoneal metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed gastric adenocarcinoma with her 2 (-), and without the history of resection of primary or metastatic lesion;
2. Peritoneal metastases from gastric cancer requiring definitive diagnosis by laparoscopy, and without gastric outflow tract obstruction and intestinal obstruction; Written (signed) informed consent;
3. Claudin 18.2 positive (≥ 25%, and the proportion of positive cells greater than 50% of the cases accounted for not less than 70%);
4. Age ≥ 18 years at registration;
5. Eastern Cooperative Oncology Group (ECOG) score ≤ 1;
6. Expected life expectancy > 3 months;
7. At least one measurable lesion, according to RECIST v1.1 as assessed by the investigator.
8. Adequate bone marrow, liver, and renal functions.

Exclusion Criteria:

1. Confirmed of evidence of distant metastasis other than peritoneal metastasis (e.g.liver metastasis, lung metastasis, para-aortic lymph node metastasis, etc.);
2. During pregnancy, within 28 days of post parturition, or during lactation;
3. Previously received immunotherapy such as PD-1/PD-L1 and CTLA-4 or targeted therapy such as Claudin 18.2.
4. Synchronous or metachronous (within 5 years) malignancies.
5. Severe mental disease, uncontrolled epilepsy, or central nervous system disease;
6. Clinically severe (i.e. active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) class II or more severe congestive heart failure or arrhythmia requiring drug intervention, or a history of myocardial infarction in the last 12 months;
7. Upper gastrointestinal obstruction or abnormal physiological function or malabsorption syndrome may affect S-1 absorbers;
8. Known peripheral neuropathy (> NCI-CTC AE 1). However, patients with only disappearance of deep tendon reflex (DTR) need not be excluded;
9. Patients on steroid or immunosuppressant treatment after organ transplant;
10. Patients with severe uncontrolled recurrent infections or other severe uncontrolled concomitant disease;
11. Moderate or severe renal damage [creatinine clearance ≤ 50 ml/min], or serum creatinine > upper limit of normal (ULN), 115 μmol/L;
12. Known dihydropyrimidine dehydrogenase (DPD) deficiency;
13. Anaphylaxis to paclitaxel or any research drug ingredient.
14. Active autoimmune disease or history of refractory autoimmune disease;
15. Subjects with hypothyroidism requiring only hormone replacement therapy and skin diseases without systemic treatment (such as vitiligo, psoriasis or alopecia) can be selected;
16. HIV antibody positive, active hepatitis B or C (hepatitis B: HBsAg positive and HBV DNA ≥10 copies/ml; hepatitis C: HCV antibody and HCV-RNA positive, requiring antiviral treatment at the same time);
17. Steroid or other systemic immunosuppressive therapy was used 14 days before admission, excluding local or physiological doses of systemic glucocorticoids (eg. no more than 10mg/day of prednisone or other glucocorticoids of equivalent dose) by nasal spray, inhalation or other routes, or hormones used to prevent allergy of contrast agents;
18. Uncontrolled arrhythmia and myocardial infarction within 12 months before admission or active tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | up to 24 months

SECONDARY OUTCOMES:
treatment related adverse events | 24 months
1-year survival rate | 12 months
Duration of Response | up to 24 months
  Duration of Response
Progressive free survival (PFS) | up to 36 months
Overall survival (OS) | up to 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Huangpu District, China

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol